CLINICAL TRIAL: NCT06895135
Title: Comparison of Efficacy of Amoxicillin Plus Clavulanic Acid and Amoxicillin in Children with Acute Otitis Media
Brief Title: Comparison of Amoxicillin and Amoxicillin + Clavulanic Acid in Treating Acute Otitis Media in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Arslan, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp130
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amoxicillin Treatment Group (Active Comparator): Participants in this arm will receive oral amoxicillin at a dose of 30mg/kg/day. They will be monitored for the resolution of symptoms, treatment failure, recurrence, and potential side effects over the course of the study.
  Interventions: Other: Amoxicillin
- Amoxicillin + Clavulanic Acid Treatment Group (Active Comparator): Participants in this arm will receive oral amoxicillin combined with clavulanic acid at a dose of 30mg/kg/day. Like the other group, they will be monitored for symptom resolution, treatment failure, recurrence, and side effects throughout the study.
  Interventions: Other: Amoxicillin; Other: Clavulanic Acid

INTERVENTIONS:
Other: Amoxicillin — Participants in this group will receive oral amoxicillin at a dosage of 30mg/kg/day. The treatment will be administered in divided doses for the duration of the study, with the aim of resolving symptoms of acute otitis media in children.
Other: Clavulanic Acid — Participants in this group will receive a combination of oral amoxicillin and clavulanic acid at a dosage of 30mg/kg/day. The medication will be given in divided doses, and participants will be monitored for symptom resolution and any potential side effects.
  Arms: Amoxicillin + Clavulanic Acid Treatment Group

SUMMARY:
This study aims to compare the effectiveness of two treatments for children with acute otitis media (middle ear infection). The two treatments being compared are amoxicillin alone and a combination of amoxicillin plus clavulanic acid. The study will help determine which treatment works better in helping children recover faster and reduce the risk of treatment failure or recurrence. By providing clearer evidence, the research aims to guide better treatment choices for children suffering from this common infection.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of two antibiotic treatments in children diagnosed with acute otitis media, a common ear infection. The two treatments being compared are amoxicillin alone and a combination of amoxicillin and clavulanic acid. Acute otitis media is a significant health concern in children, causing pain, fever, and possible hearing loss.

The study will be conducted as a randomized controlled trial at the Department of Pediatric Medicine, Nishtar Hospital, Multan. A total of 162 children, aged 1 to 5 years, will be enrolled in the study. They will be randomly assigned to one of two treatment groups: one group will receive amoxicillin, and the other group will receive amoxicillin plus clavulanic acid. The children will be monitored throughout their treatment to assess how quickly their symptoms resolve, whether they experience treatment failure or recurrence, and if they develop any side effects.

The study aims to provide clearer evidence on the efficacy of the combination treatment (amoxicillin + clavulanic acid) compared to amoxicillin alone. By analyzing treatment outcomes such as symptom resolution time, side effects, and recurrence, the study will help inform clinical decisions and improve treatment protocols for acute otitis media in pediatric patients. The data will be analyzed using statistical software to determine whether the combination therapy leads to faster recovery and fewer complications. The findings from this study will contribute to better management of upper respiratory infections in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 5 years
* Diagnosed with acute otitis media (as per operational definition)
* Both male and female participants
* Parental consent obtained

Exclusion Criteria:

* Children with allergies or contraindications to the trial drugs (amoxicillin or amoxicillin + clavulanic acid)
* Children with asthma or chronic obstructive pulmonary disease (COPD) (as per medical record)
* Children who have received treatment with the trial drugs within the past month
* Children already enrolled in other research programs or who have received trial treatment
* Children with any comorbid conditions that may interfere with the study

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time to Symptom Resolution (in Days) | From enrollment to the resolution of symptoms, assessed daily until symptoms are resolved, up to a maximum of 4 weeks.
  How Measured: The number of days it takes for the symptoms of acute otitis media (fever, ear pain, bulging tympanic membrane) to completely resolve after starting treatment will be recorded. Participants will be assessed daily until the resolution of symptoms. The assessment will be made by the treating physician based on clinical signs observed through otoscopy and patient-reported outcomes (such as pain relief).
  Criteria for Resolution: Symptoms are considered resolved when the child no longer experiences ear pain, fever, or any other signs of infection. The tympanic membrane will appear normal during otoscopy, with no visible bulging or signs of fluid accumulation.
Number of Participants with Treatment Failure | Assessed at 4 weeks from the start of treatment.
  Treatment failure is defined as the failure to resolve symptoms within 4 weeks of starting treatment. If symptoms persist or worsen despite the antibiotic treatment, the physician will classify the case as treatment failure and change the antibiotic regimen.

IPD SHARING:
Plan to Share IPD: Undecided